CLINICAL TRIAL: NCT07293910
Title: Safety and Efficacy of Vonoprazan vs Proton Pump Inhibitor With Vitamin D or Probiotics Based Triple Therapy for Eradication of Helicobacter Pylori Infection
Brief Title: Vonoprazan vs Proton Pump Inhibitor With Vitamin D or Probiotics Based Triple Therapy for Eradication of Helicobacter Pylori Infection
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hagar Khaled Bassuony Dewidar, Assistant Lecturer of Clinical Pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Helicobacter Pylori
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: HELICOBACTER PYLORI INFECTIONS; Helicobacter Infection; Helicobacter Pylori Gastrointestinal Tract Infection; Helicobacter Pylori Infected Patients
Keywords: Helicobacter Pylori; Vonoprazan; Vitamin D; Probiotics; Lactobacillus; C-reactive protein; Tumor necrosis factor alpha; Malondialdehyde
MeSH Terms: conditions — Helicobacter Infections | interventions — Vitamin D; Probiotics; Amoxicillin; Clarithromycin; Proton Pump Inhibitors; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vonoprazan group (Active Comparator): 22 patients will receive vonoprazan (20 mg) with amoxicillin (1000 mg) and clarithromycin (500 mg) twice daily for 2 weeks
  Interventions: Drug: Vonoparazan; Drug: Amoxicillin; Drug: Clarithromycin 500 mg
- Probiotic group (Active Comparator): 22 patients will receive proton pump inhibitor-based triple therapy omeprazole /pantoprazole (40 mg) with amoxicillin (1000 mg) and clarithromycin (500 mg) twice daily with lactobacillus acidophilus (5 billion CFU) three times daily for 2 weeks.
  Interventions: Drug: Probiotic; Drug: Amoxicillin; Drug: Clarithromycin 500 mg; Drug: Proton Pump Inhibitor (PPI) Therapy
- Vitamin D group (Active Comparator): 22 patients will receive proton pump inhibitor-based triple therapy omeprazole /pantoprazole (40mg) with amoxicillin (1000 mg) and clarithromycin (500 mg) twice daily with vitamin D (2000 I.U.) once daily for 2 weeks.
  Interventions: Drug: Vitamin D; Drug: Amoxicillin; Drug: Clarithromycin 500 mg; Drug: Proton Pump Inhibitor (PPI) Therapy

INTERVENTIONS:
Drug: Vonoparazan — Vonoprazan: Potassium competitive acid blocker
  Arms: Vonoprazan group
Drug: Vitamin D — MIcronutrient
  Arms: Vitamin D group
Drug: Probiotic — Lactobacillus acidophilus
  Arms: Probiotic group
Drug: Amoxicillin — Amoxicillin is penicillin-type antibiotic used to treat a wide range of bacterial infections.
Drug: Clarithromycin 500 mg — Clarithromycin is a prescription macrolide antibiotic used to treat a variety of bacterial infections
Drug: Proton Pump Inhibitor (PPI) Therapy — Proton Pump Inhibitors (PPIs) are powerful medications that significantly reduce stomach acid production by blocking the H+/K+ ATPase enzymes (proton pumps) in the stomach lining,
  Arms: Probiotic group; Vitamin D group

SUMMARY:
Helicobacter pylori is a Gram-negative, spiral-shaped bacterium that infects up to 50% of the world's population, residing in the gastric mucosa and using the mucus layer for protection from the stomach's high acidity. Its clinical significance is profound: it is classified as a Group 1 carcinogen by the World Health Organization and is a primary cause of chronic gastritis, peptic ulcers, gastric lymphoma, and gastric carcinoma. The current first-line treatment, a PPI-based triple therapy (PPI + clarithromycin + amoxicillin), is experiencing a decline in efficacy (cure rates of 50-70%) due to widespread antibiotic resistance and compliance issues. To overcome this, newer agents like Vonoprazan Fumarate, a Potassium-Competitive Acid Blocker (P-CAB), are being adopted. Vonoprazan works by reversibly inhibiting the H+, K+ ATPase pump achieving stronger and longer-lasting acid suppression than PPIs because it does not require acid activation and is more stable in an acidic environment. In addition to pharmacological treatment, adjunctive therapies show promise. Vitamin D, acting through Vitamin D Receptor (VDR), assists in eradication by upregulating antimicrobial proteins like beta-defensin and cathelicidin, and its metabolite can cause bacterial cell lysis. Probiotics (primarily Lactobacillus and Bifidobacterium strains) enhance eradication rates by restricting bacterial growth, inhibiting adhesion, and exerting an anti-inflammatory effect through decreased interleukin-8 production. Finally, helicobacter pylori infection is marked by significant inflammation and oxidative stress. The bacterial protein TIP alpha induces high levels of the pro-inflammatory cytokine TNF alpha. Furthermore, the infection increases free radical production, leading to oxidative stress reflected by high levels of malondialdehyde. Systemic inflammation is also evident as helicobacter pylori infection is associated with significantly elevated serum C-reactive protein levels, which decrease upon successful eradication.

Aim of the work:

This study aims at evaluating the safety and efficacy of Vonoprazan vs Proton Pump Inhibitor with Vitamin D or Probiotics Based Triple Therapy for Eradication of Helicobacter Pylori Infection.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) is a gram-negative spiral-shaped bacterium that affects up to 50% of the population worldwide, with a higher prevalence in developing countries. H. pylori is found primarily in the human gastric mucosa, its natural habitat, where it remains close to epithelial cells. H. pylori is attracted to the gastric mucus layer, which offers cover and protection from the high acidity in the stomach and promotes better cell motility.

It has been identified as a group 1 carcinogen by the world health organization (WHO) and is associated with the development of gastric cancer. It is also the most important cause for chronic or atrophic gastritis, peptic ulcer, gastric lymphoma, and gastric carcinoma.

First-line therapy for the treatment of H. pylori infection is a triple therapy consisting of a clarithromycin antibiotic, amoxicillin and proton pump inhibitor (PPI). PPI-based triple therapy has been described to be losing its efficacy against H. pylori, with eradication cure rates ranging as low as 50 to 70%, due to high rates of antibiotic resistance, high rates of antibiotic-associated side effects, and weak compliance. Vonoprazan fumarate is a potassium-competitive acid blocker (P-CAB), which is agent that inhibits H+ ,K+ adenosine triphosphatase (ATPase) through reversible K+ competitive ionic binding that results in the inhibition of gastric acid secretion. Because vonoprazan has a relatively high pKa value and is stable in an acidic environment, it can accumulate in the acidic compartment of gastric parietal cells, unlike PPIs. In addition, vonoprazan does not require acid activation, in contrast to PPIs. Thus, vonoprazan can achieve stronger, longer-lasting suppression of gastric acid secretion than PPIs can. Murakami et al. compared the H. pylori eradication rate of vonoprazan with that of PPIs for patients with gastroduodenal ulcers in a randomized, double-blind,multicenter, parallel-group comparative study. The results demonstrated superiority of vonoprazan to lansoprazole regarding the therapeutic effect on H. pylori eradication.

Vitamin D is a micronutrient that regulates bone metabolism. Through vitamin D receptor (VDR), vitamin D plays biological activities. Several studies have uncovered the relationship between vitamin D and H pylori infection, and vitamin D and H pylori eradication. A previous study reported that infected macrophages upregulate the production of β-defensin to kill H pylori strains by VDR. Vitamin D3 can also induce the VDR- cathelicidin antimicrobial protein (CAMP) signaling pathway to eradicate H. pylori in the stomach. Several studies have found that vitamin D3 decomposition product 1 (VDP1) can induce cell membrane collapse, leading to the lysis of H. pylori cells.

Probiotics refer to a group of beneficial bacteria which are gaining acceptance in improving the eradication rate of H. pylori by restricting its growth (anti-microbial activity) and inhibiting subsequent inflammatory processes related to H. pylori infection. Antimicrobial activity is mainly through inhibition of H. pylori adhesion and invasion of gastric epithelial cells and anti-inflammatory role through decreasing interleukin-8 production. The majority of probiotics are of the genera, Lactobacillus and Bifidobacterium. Both strains mostly possess properties of acid tolerance and antimicrobial activity. It was reported that the eradication rate was higher in patients who received probiotics with standard therapy compared to those patients treated with standard therapy alone. A specific H. pylori protein, tumor necrosis factor alpha (TNF-α)-inducing protein (Tipα), plays a significant role by directly inducing TNF-α and other pro-inflammatory cytokines which contributes to gastritis, peptic ulcers, and gastric cancer. TNF-α level is reported to be higher in individuals infected with H. pylori in comparison to uninfected individuals.

H. pylori increases free radicals production which leads to oxidative stress and can involve DNA and gastric tissue damage. It was reported that malondialdehyde (MDA) levels are significantly higher in H. pylori-infected gastric mucosa, compared to normal tissue, and the levels of MDA are significantly decreased after H. pylori eradication. C-reactive protein (CRP) is an acute-phase inflammatory liver protein, it facilitates the recognition of foreign pathogens and the phospholipid constituents of damaged cells. It was reported that CRP serum levels were significantly elevated in H. pylori-infected patients and significantly decreased after H. pylori eradication.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients. • Patients ≥ 18 and <80 years old.

Patients with confirmed diagnosis of H. pylori infection using either stool antigen test, urea breath test or endoscopy.

Exclusion Criteria:

* Pregnant or lactating patients. • Patients with inflammatory diseases. • Patients sensitive to any of the regimens' components. • Patients who had received a previous eradication therapy, recent use of antimicrobial agents, proton pump inhibitors, and H2 receptor blockers within 1 month.

Patients with previous incidents of gastric or duodenal bleeding, gastric surgery or gastric malignancy.

• Patients with active liver disease.

• Patients with renal impairment.

• Concurrent use of liver enzyme inducers, inhibitors or drugs with high plasma protein binding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Detection of H pylori eradication difference among the three groups through stool antigen test 4 weeks after completion of therapy. | 4 weeks after completion of therapy
  We will asses the presence or absence of H pylori through fecal antigen test four weeks after completion of therapy among the three groups It will be assessed as either positive or negative

SECONDARY OUTCOMES:
Changes in serum levels of the measured biological markers | 4 weeks after completion of therapy
  The secondary outcome is the changes in serum levels of TNF-alpha, C-reactive protein and Malondialdehyde 4 weeks after completion of therapy
Change in Gastrointestinal Symptom Rating Scale Questionnaire total score from baseline to completion of therapy and 4 weeks after completion of therapy | From baseline to completion of therapy and 4 weeks after completion of therapy
  change in Gastrointestinal Symptom Rating Scale Questionnaire total score from baseline to completion of therapy and 4 weeks after completion of therapy as it is a validated, 15-item questionnaire used to assess GI symptom severity, grouping symptoms into five clusters: Reflux, Abdominal Pain, Indigestion, Diarrhea, and Constipation, scored on a 1-7 Likert scale (1=no discomfort, 7=very severe).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gombart AF, Borregaard N, Koeffler HP. Human cathelicidin antimicrobial peptide (CAMP) gene is a direct target of the vitamin D receptor and is strongly up-regulated in myeloid cells by 1,25-dihydroxyvitamin D3. FASEB J. 2005 Jul;19(9):1067-77. doi: 10.1096/fj.04-3284com. PMID 15985530
- [Background] Wanibuchi K, Hosoda K, Ihara M, Tajiri K, Sakai Y, Masui H, Takahashi T, Hirai Y, Shimomura H. Indene Compounds Synthetically Derived from Vitamin D Have Selective Antibacterial Action on Helicobacter pylori. Lipids. 2018 Apr;53(4):393-401. doi: 10.1002/lipd.12043. Epub 2018 May 16. PMID 29766504
- [Background] Murakami K, Sakurai Y, Shiino M, Funao N, Nishimura A, Asaka M. Vonoprazan, a novel potassium-competitive acid blocker, as a component of first-line and second-line triple therapy for Helicobacter pylori eradication: a phase III, randomised, double-blind study. Gut. 2016 Sep;65(9):1439-46. doi: 10.1136/gutjnl-2015-311304. Epub 2016 Mar 2. PMID 26935876
- [Background] Hori Y, Imanishi A, Matsukawa J, Tsukimi Y, Nishida H, Arikawa Y, Hirase K, Kajino M, Inatomi N. 1-[5-(2-Fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl]-N-methylmethanamine monofumarate (TAK-438), a novel and potent potassium-competitive acid blocker for the treatment of acid-related diseases. J Pharmacol Exp Ther. 2010 Oct;335(1):231-8. doi: 10.1124/jpet.110.170274. Epub 2010 Jul 12. PMID 20624992
- [Background] Iannone A, Giorgio F, Russo F, Riezzo G, Girardi B, Pricci M, Palmer SC, Barone M, Principi M, Strippoli GF, Di Leo A, Ierardi E. New fecal test for non-invasive Helicobacter pylori detection: A diagnostic accuracy study. World J Gastroenterol. 2018 Jul 21;24(27):3021-3029. doi: 10.3748/wjg.v24.i27.3021. PMID 30038469
- [Background] Schreiber S, Konradt M, Groll C, Scheid P, Hanauer G, Werling HO, Josenhans C, Suerbaum S. The spatial orientation of Helicobacter pylori in the gastric mucus. Proc Natl Acad Sci U S A. 2004 Apr 6;101(14):5024-9. doi: 10.1073/pnas.0308386101. Epub 2004 Mar 25. PMID 15044704
- [Background] Ceylan A, Kirimi E, Tuncer O, Turkdogan K, Ariyuca S, Ceylan N. Prevalence of Helicobacter pylori in children and their family members in a district in Turkey. J Health Popul Nutr. 2007 Dec;25(4):422-7. PMID 18402185